CLINICAL TRIAL: NCT04675255
Title: WU 360: Assessing the Impact of Integrase Strand Transfer Inhibitors (INSTI) to Protease Inhibitor (PI) Switch on Insulin Sensitivity and Fat Metabolism (ADIPOSITY): a Sub-study of DEFINE
Brief Title: Assessing the Impact of INSTI to PI Switch on Insulin Sensitivity and Fat Metabolism
Acronym: ADIPOSITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202008043
Record Dates: First submitted 2020-10-13; First posted 2020-12-19 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: HIV I Infection; Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate switch (Active Comparator): Immediate switch
  Interventions: Procedure: Frequently sampled glucose tolerance testing; Procedure: abdominal subcutaneous adipose tissue biopsy; Procedure: MRI scan to assess intrahepatic triglyceride content
- Delayed switch (Active Comparator): Delayed switch
  Interventions: Procedure: Frequently sampled glucose tolerance testing; Procedure: abdominal subcutaneous adipose tissue biopsy; Procedure: MRI scan to assess intrahepatic triglyceride content

INTERVENTIONS:
Procedure: Frequently sampled glucose tolerance testing — Frequently sampled glucose tolerance testing
Procedure: abdominal subcutaneous adipose tissue biopsy — abdominal subcutaneous adipose tissue biopsy
Procedure: MRI scan to assess intrahepatic triglyceride content — MRI scan to assess intrahepatic triglyceride content

SUMMARY:
A substudy of TMC114FD2HTX4004 that will perform glucose tolerance testing, adipose testing and MRI scan at baseline, 12 and 24 weeks post switch of ART medications.

DETAILED DESCRIPTION:
Synopsis Full study title: Assessing the impact of integrase strand transfer inhibitors (INSTI) to protease inhibitor (PI) switch on insulin sensitivity and fat metabolism (ADIPOSITY): a sub-study of DEFINE

Endpoints and objectives:

The following endpoints will be determined 12 and 24 weeks after switch from an INSTI-based antiretroviral therapy (ART) regimen to a PI-based regimen:

Primary endpoint: Change in insulin sensitivity (SI) at 12 weeks assessed by using a 3-hour frequently sampled oral glucose tolerance testing (fsOGTT).

Secondary endpoints: 1) Change in insulin sensitivity (SI) at 24 weeks assessed by using a 3-hour frequently sampled oral glucose tolerance testing (fsOGTT); 2) Change in insulin secretion during the fsOGTT assessed by using C-peptide deconvolution; 3) Change in intrahepatic triglyceride (IHTG) content measured by magnetic resonance imaging (MRI); 4) Change in adipocyte size by the osmium tetroxide fixation technique; and 5) Change in expression of genes associated with adipose tissue development, lipogenesis, inflammation and endocrine function by RNA sequencing.

Hypothesis: Insulin sensitivity will improve following switch from INSTIs to PIs

ELIGIBILITY:
Inclusion Criteria:

* • Must be enrolled in the DEFINE study TMC114FD2HTX4004

  * Must sign an ICF indicating that they understand the purpose of, and procedures required for, the study and are willing to participate in the study.

Exclusion Criteria:

* • Contraindication to magnetic resonance imaging as determined by institutional policy.

  * Current diagnosis of diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity measured by homeostatic model assessment for insulin resistance {HOMA_IR} | 12 weeks
  Change in insulin sensitivity (SI) at 12 weeks assessed by using a 3-hour frequently sampled oral glucose tolerance testing (fsOGTT).to calculate HOMA_IR

SECONDARY OUTCOMES:
Intrahepatic triglyceride (IHTG) content measure by magnetic resonance | 12 weeks
  Change in intrahepatic triglyceride (IHTG) content measured by magnetic resonance imaging (MRI
Intrahepatic triglyceride (IHTG) content measure by magnetic resonance | 24 weeks
  Change in intrahepatic triglyceride (IHTG) content measured by magnetic resonance imaging (MRI
Adipocyte size measured by osmium tetroxide fixation technique | 12 weeks
  Change in adipocyte size by the osmium tetroxide fixation technique
Adipocyte size measured by osmium tetroxide fixation technique | 24 weeks
  Change in adipocyte size by the osmium tetroxide fixation technique
Adipocyte gene expression correlated with adipose tissue development | 12 weeks
  Change in expression of adipose tissue genes correlated with adipose tissue development, lipogenesis, inflammation and endocrine function measured by RNA sequencing
Adipocyte gene expression correlated with adipose tissue development | 24 weeks
  Change in expression of adipose tissue genes correlated with adipose tissue development, lipogenesis, inflammation and endocrine function measured by RNA sequencing
Insulin Sensitivity measured by homeostatic model assessment for insulin resistance {HOMA_IR} | 24 weeks
  Change in insulin sensitivity (SI) at 12 weeks assessed by using a 3-hour frequently sampled oral glucose tolerance testing (fsOGTT).to calculate HOMA_IR

CONTACTS AND LOCATIONS:
Overall Officials: Jane O'Halloran, MB BA PhD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan